CLINICAL TRIAL: NCT00674245
Title: The Effect Of Pantoprazole 40 mg Once Daily Versus Placebo On The Power Spectral Analysis Of The Sleep Electroencephalogram (EEG) Of Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: Effect of Pantoprazole 40mg Daily vs Placebo on Power Spectral Analysis of the Sleep EEG of Patients With GERD.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Southern Arizona VA Health Care System (U.S. Federal Agency)
Responsible Party: Ronnie Fass, MD, Southern Arizona VA Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0001-01 & R&D#00-77
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: heartburn; acid reflux; GERD; spectrum analysis; electroencephalogram; esophagitis; peptic
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Esophagitis | interventions — Pantoprazole; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pantoprazole (Active Comparator): 40 mg once daily for four weeks improves sleep quality in patients with GERD
  Interventions: Drug: Pantoprazole
- placebo (Placebo Comparator): To determine if treatment with pantoprazole 40 mg once daily vs placebo improves sleep outcome in patients with GERD.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pantoprazole — 40 mg once daily for 4 weeks
  Other Names: Protonix; PPI
  Arms: Pantoprazole
Drug: Pantoprazole — 40 mg once daily improves sleep quality in patients with GERD.
  Other Names: Protonix; PPI
  Arms: Pantoprazole
Drug: placebo — 40 mg once daily for 4 weeks
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
The purpose of this research study is to determine if treatment with pantoprazole 40 mg daily versus a placebo improves sleep quality in patients with gastroesophageal reflux disease (GERD). Another purpose is to determine if treatment with pantoprazole 40 mg once daily versus a placebo improves sleep outcomes in patients with gastroesophageal reflux disease using spectral analysis of sleep electroencephalogram (EEG).

DETAILED DESCRIPTION:
It appears that the presence of intraesophageal stimuli alone may not be sufficient to elicit symptoms of heartburn. Most acid reflux events (>80%-90%) do not reach conscious level and thus are not perceived.[3] It is yet to be determined what factors enhance our perception of esophageal stimuli and may help to elevate them to the conscious level. In recent years, central and peripheral factors that may enhance our perception of intraesophageal stimuli have been evaluated. Intraduodenal fat infusion was shown to enhance perception of intraesophageal acid in patients with GERD.[4] This study suggested that fat is an important modulator of postprandial GERD symptoms. Central factors, such as stress and psychological comorbidity, also appear to have an important role in symptom generation in patients with GERD, regardless if esophageal inflammation is present or absent.[5-8] Thus, by modulating brain-gut interactions, perception of pathological and probably physiological events in the esophagus of patients with GERD may be altered.

Poor sleep is a central factor that may enhance perception of intraesophageal stimuli and thus elevate them to the conscious level. Several studies have demonstrated that patients with fibromyalgia or irritable bowel syndrome report increased symptoms due to sleep abnormalities.[9, 10] Similar reports in patients with GERD are not available. A subset of patients with GERD experience nocturnal heartburn that may awaken them during the night. In others, despite lack of nocturnal symptoms, sleep abnormalities may occur due to acid reflux events. In both cases, GERD leads to poor sleep, and that in turn may enhance perception of intraesophageal stimuli, leading to reports of increased frequency and severity of perceived GERD symptoms. Thus, poor sleep may be a crucial factor in symptom generation and exacerbation of patients with GERD.

Recently, we have used a novel technique, power spectral analysis of the sleep electroencephalogram (EEG), to assess patients with heartburn and erosive esophagitis and those with heartburn but without erosive esophagitis.[11] We were able to show that among heartburn patients with GERD, EEG spectral power during sleep is shifted towards higher frequencies as compared to heartburn patients without GERD despite similar sleep architecture.

Several recent therapeutic trials in GERD patients have failed to demonstrate improvement in polysomnographic studies despite improvement in GERD-related symptoms and subjective reports of sleep quality.[12] Spectral analysis of the sleep EEG might be a more sensitive tool than polysomnographic study in assessing objective improvement of sleep in patients receiving antireflux treatment.

In summary, sleep disturbances in patients with GERD are poorly recognized and rarely elicited during clinic visits despite their significant impact on patients' quality of life and probably perception of disease severity. Several studies have demonstrated improvement of subjective reports of sleep quality in patients with GERD receiving antireflux treatment. However, the effect of potent antireflux therapy on objective sleep parameters has yet to be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 yrs of age
* 2 to 3 episodes of GERD/week
* erosive esophagitis or abnormal 24 hr pH
* able to read and understand, complete questionnaires

Exclusion Criteria:

* barrett's esophagus or peptic stricture on endoscopy
* normal EGD and normal 24 hour pH
* previous upper GI surgery
* comorbidity (cardiovascular, respiratory, renal, hepatic)
* use of narcotics or pain medication on regular basis
* insomnia, shift work sleep disorder, sleep apnea, restless leg syndrome
* diabetes, scleroderma or neuromuscular disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Symptom control after 4 weeks of treatment. | April 2008 to July 2010
  To determine if treatment with pantoprazole 40 mg daily vs placebo improves sleep quality in patients with GERD.

SECONDARY OUTCOMES:
Effect of Pantoprazole 40 mg Daily vs Placebo on the Power Spectral Analysis of the Sleep Electroencephalogram of Patients With GERD. | April 2008-July 2010
  To determine if treatment with pantoprazole 40 mg once daily vs placebo improves sleep outcome in patients with GERD using spectral analysis of sleep electroencephalogram.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — Southern VA Health Care System
Locations (1):
- Southern Arizona VA Health Care System, Tucson, Arizona, United States

REFERENCES:
- [Background] Fass R, Fullerton S, Tung S, Mayer EA. Sleep disturbances in clinic patients with functional bowel disorders. Am J Gastroenterol. 2000 May;95(5):1195-2000. doi: 10.1111/j.1572-0241.2000.02009.x. PMID 10811327
- [Background] Wiklund IK, Junghard O, Grace E, Talley NJ, Kamm M, Veldhuyzen van Zanten S, Pare P, Chiba N, Leddin DS, Bigard MA, Colin R, Schoenfeld P. Quality of Life in Reflux and Dyspepsia patients. Psychometric documentation of a new disease-specific questionnaire (QOLRAD). Eur J Surg Suppl. 1998;(583):41-9. PMID 10027672
- [Background] Orr WC, Goodrich S, Robert J. The effect of acid suppression on sleep patterns and sleep-related gastro-oesophageal reflux. Aliment Pharmacol Ther. 2005 Jan 15;21(2):103-8. doi: 10.1111/j.1365-2036.2005.02310.x. PMID 15679759
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956
- [Background] Goldsmith G, Levin JS. Effect of sleep quality on symptoms of irritable bowel syndrome. Dig Dis Sci. 1993 Oct;38(10):1809-14. doi: 10.1007/BF01296103. PMID 8404401